A Randomized Clinical Trial of BaDuanJin in Treatment of Attention Deficit Hyperactivity Disorder with Hyperactive-Impulsive Symptom

# STATISTICAL ANALYSIS PLAN

Clinicaltrials.gov Number: NCT04282460

Protocol vision and data: Vision 1.0 September 27, 2021

# Core writing group

| Role | Researcher Name | |
|--------------------|-----------------|------------|
| Chief investigator | Daqian Zhu | Dayson Thu |
| Trial statistician | Weili Yan | Weili You |
| Trial statistician | Yin Wang | Vin INMA |

# SAP version history

Chief investigator: Phd Daqian Zhu

Trial statisticians: Prof Weili Yan; Phd Yin Wang

SAP authors: Prof Weili Yan; Yin Wang; Mengyao Li; Yu Li

| Version Date | SAP version# | Details of Changes | Signatures |
|---|---|---|---|
| September 27, 2021 | 1.0 | - | - |
| December 8, 2021 | 1.2 | Adding detail description of multiple imputations | Weilyon<br>Win Wans |
| December 12, 2021 | 1.3 | Add Graphical/Table displays | Dagranzking wan |
| July 26, 2022 | 1.4 | Adding more secondary outcomes (CANTAB test and BRIEF2 scale) analyses; Adding effect size description | Dargven Whi<br>Weilifon |
| October 25, 2022 | 2.0 | Adding more detail information of sample size calculation; Adding detail description of GLMM estimation | Vin Wang<br>Defron when<br>Weelifor |

Protocol A Randomized Clinical Trial of BaDuanJin in Treatment of Attention Deficit Hyperactivity Disorder with Hyperactive-Impulsive Symptom

# Statistical Analysis plan

The Data Management and Statistical Analysis Plan is directed to support the aims of the study

Version 2.0

September 27, 2021 Draft

October 25, 2022 Modified

Yin Wang Weili Yan

#### Statistical Analysis Plan

| Intro | oduction | 2 |
|---|---|---|
| 1. | Study Objective and Outcomes | 2 |
| | 1.1. Study Objective | 2 |
| | 2.2. Outcomes | 2 |
| | 2.2.1. Primary outcome | 2 |
| | 2.2.2. Secondary outcomes | 3 |
| 3. St | udy Design | 4 |
| | 3.1. Design | 4 |
| | 3.2. Trial Sites | 5 |
| | 3.3. Interventions | 5 |
| | 3.3.1. Experimental group: | 5 |
| | 3.3.2. Control group: | 5 |
| | 3.4. Randomization | 5 |
| | 3.5. Blinding | 6 |
| | 3.6. Sample Size | 6 |
| 4.Aı | nalysis Consideration | 7 |
| | 4.1. Trial hypothesis | 7 |
| | 4.2. Study population data sets | 7 |
| | 4.3. Study Close Date | 8 |
| | 4.4. Data Cleaning | 8 |
| | 4.5. Data Check-up. | 8 |
| 5. St | atistical Analyses | 8 |
| | 5.1. Primary Outcome Analysis | 8 |
| | 5.1.1. ITT analysis of the primary outcome - the primary analysis | 8 |
| | 5.1.2. Per-protocol analyses of the primary outcome | 9 |
| | 5.1.3. Covariate adjusted analysis of the primary outcome | 9 |
| | 5.1.4. Subgroup analyses of the primary outcome | 9 |
| | 5.2. Secondary Outcome Analysis | .10 |
| | 5.2.1. Handling of Missing data | .10 |
| 6.Ge | eneral Considerations for Data Analyses | |
| | 6.1. Other Data Summaries | .11 |
| | 6.2. Graphical/Table Displays | |
| 7.St | udy variable list | .18 |
| 8 Re | eference | 26 |

# Introduction

ADHD is a common neurodevelopmental disorder characterized by a persistent pattern of inattention and/or hyperactivity and impulsivity, resulting in functional impairment in multiple settings. The prevalence in China is estimated to be 6.26%[1]. Physical exercise is indicted as an alternative approach to the treatment of ADHD, used independently or complementary to medication or behavioral interventions that can yield both acute and lasting positive effects on executive function, which is known as the core neurobiological deficit in ADHD. Baduanjin exercise, a combination of physical exercise and Chinese qigong movement, is considered as a potential alternative treatment to ADHD in Traditional Chinese Medicine (TCM). This study aims to evaluate the effectiveness of Baduanjin exercise on reducing the hyperactive-impulsive symptoms of children with ADHD compared with the current treatment, routine exercise, as the control treatment.

# 1. Study Objective and Outcomes

# 1.1. Study Objective

The aim of this randomized controlled trial is to explore the effectiveness of Baduanjin practice versus routine physical exercise in improving Hyperactive-Impulsive Symptoms among pediatric ADHD patients.

#### 2.2. Outcomes

# 2.2.1. Primary outcome

Hyperactivity/Impulsivity score change assessed by doctor version of SNAP-IV scale at 3th month.

Time Frame: Baseline, 3th month after initiation of intervention

Type: repeated measured continuous variable

### 2.2.2. Secondary outcomes

(1) Hyperactivity/Impulsivity score change assessed by doctor version of SNAP-IV scale at 6th month.

Time Frame: Baseline, 6th month after initiation of intervention

Type: repeated measured continuous variable

(2) Hyperactivity/Impulsivity score changes assessed by parent version of SNAP-IV scale.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(3) Changes of Scoring evaluation of the TCM symptoms.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(4) Change scores of inattention and Oppositional Defiant Disorder (ODD) subscale assessed by doctor version of SNAP-IV scale.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(5) Change scores of inattention and Oppositional Defiant Disorder (ODD) subscale score assessed by parent version of SNAP-IV scale.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(6) The changes of Weiss Functional Impairment Rating Scale (WFIRS) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(7) The changes of parent version of Achenbach Child Behavior Checklist (CBCL) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(8) The changes of Child version of Achenbach Child Behavior Checklist (CBCL) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(9) The changes of CANTAB test (neuropsychological tests) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(10) The changes of BRIEF2 scale (ecological rating scale) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(11) The changes of Visual Perception-2nd edition (DTVP-2) score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

(12) The changes of Child Sensory Integration Checklist score.

Time Frame: Baseline, 3th month and 6th month after initiation of intervention

Type: repeated measured continuous variable

# 3. Study Design

# 3.1. Design

The trial is a single-blind, superiority, randomized controlled trial. Patients fulfil the eligibility criteria as outlined in the protocol are invited to participate consecutively and are randomized individually to control or experimental arm. Block randomization (block size of 4) will be applied.

Statistical Analysis Plan

3.2. Trial Sites

Single center: Children's hospital of Fudan University

Children's Hospital of Fudan University is a comprehensive tertiary pediatric hospital

and one of the national children's medical centers. Patients are enlisted at the clinic of

both Child psychology department and TCM department.

3.3. Interventions

3.3.1. Experimental group

Intervention: Baduanjin exercise

Use the Baduanjin training system to practice the whole set of Baduanjin at least once

a day and at least 5 days each week and last for 3 months.

More detailed information of Baduanjin practice is presented in the protocol.

3.3.2. Control group

Active Comparator: Regular physical exercise

Take routine physical exercise (any kind of routine physical exercise including jogging,

bike-riding, badminton, table tennis, soccer, basketball, aerobics and rope skipping.)

for 30 minutes, 5 days each week under the supervision of caregivers in addition to

regular physical activities at school and last for 3 months.

3.4. Randomization

According to the random seeds (seed:20200618), numbers from 1 to 6 were randomly

generated by the R software (version 4.0.0) for each block, and each number

corresponded to one of six plans for allocating four participants of the block to two

arms in a 1:1 ratio. Each allocation sequence was placed in small, opaque, and sealed

envelopes numbered and marked in order from one to four and were enclosed in a larger,

opaque, and sealed envelope marked with the block number.

A randomization plan and concealed envelopes were prepared by an independent team of statisticians from the Clinical Trial Unit (CTU) of the Children's Hospital of Fudan University. Recruited patients will be randomly allocated in a 1:1 ratio to the control or experimental group based on the randomization plan: After obtaining signed informed consent from the eligible participant, the trained physician will meet with the prespecified institutional nurse to achieve the allocation plan for the very participant, as indicated by the corresponding envelope. Block envelopes and the four enclosed small envelopes will be opened in order. The nurse will administer the allocation record form in front of the physician.

## 3.5. Blinding

The physicians in charge of outcome evaluation will be blinded about the grouping of the patients. The trial statistician will also be blinded regarding the treatment code when he develops the statistical analysis plan and writes the statistical programs, which will be validated and completed using dummy randomization codes. The actual allocation will only be provided to the study team after lock of the database.

## 3.6. Sample Size

The sample size was calculated based on the primary outcome. According to our 3 months pilot study, the change score of Hyperactivity/Impulsivity assessed by doctor version of SNAP-IV scale in Baduanjin practice group (N=23) was 3.52 with a standard deviation of 5.81. Based on the outpatient data among ADHD patients, the mean change score Hyperactivity/Impulsivity assessed by doctor version of SNAP-IV scale in regular physical exercise patients was 0.37 with a standard deviation of 3.72. We assumed that the difference in the mean change score between Baduanjin practice group and regular

physical exercise group was 3.1 a standard deviation of 5.8. So as to demonstrate superiority with 80% of power and a significance level of 0.05 (two-sided), at least 56 participants for each arm will be required. With an anticipated a drop-out rate of 5%, a total of 120 participants need to be randomized.

# 4. Analysis Consideration

## 4.1. Trial hypothesis

The hypothesis H0: "No difference in the change of Hyperactivity/Impulsivity score assessed by doctor version of SNAP-IV scale at 3th month between two groups." will be tested against the alternative" H1: "The change of Hyperactivity/Impulsivity score assessed by doctor version of SNAP-IV scale at 3th month is different between two groups."

## 4.2. Study population data sets

Two study populations will be considered in the analysis as follows:

#### -Intent-to-Treat population

Intent-to-treat (ITT) population will be defined at the moment the randomization is performed. This will be the primary analysis for the trial.

Particints will be excluded from the ITT analysis if the primary outcome is missing, forming a modified ITT population (mITT).

#### -Per-protocol population

Participants will be excluded from the per-protocol population if their qualified exercise days (more than 30 minutes and the maximum heart rate during the exercise should be over 120 beats) less than 48 days. The experimental group in the per-protocol analysis will be defined according to what the participant actual receive. This population will be used for the supportive analyses.

#### -Safety population

Participants who were given any exercise-relate-treatment would be included in this population. Adverse reactions and events would be recorded. This population will be used for the supportive analyses.

## 4.3. Study Close Date

The data collection close date is the date on which the last patient completed follow-up to achieve outcomes (complete 6 months follow-up).

## 4.4. Data Cleaning

The data will then be checked to ensure that there are no erroneous entries and that all missing data is properly coded. Any changes will be made on the ACCESS database.

## 4.5. Data Check-up

Once all data have been inputted and checked, the database will be locked and a data download request made. The data will be downloaded into SAS and R for statistical analyses.

# 5. Statistical Analyses

# **5.1. Primary Outcome Analysis**

# 5.1.1. ITT analysis of the primary outcome - the primary analysis

The primary outcome is a repeated measured continuous variable, Hyperactivity/Impulsivity score change in doctor rated SNAP-IV scale. The primary analysis will be based on the mITT population as defined above. Generalized liner

mixed model (GLMM) will be performed using maximum likelihood (ML) method with treatment (binary) and time (ordinal) and interaction of treatment with time as fixed effect, and ID as random effect. Gaussian distribution and identity link function will be used in the GLMM model. Mean difference and 95% confidence intervals (CI) between groups at each time point will be estimated based on the fitted GLMM model.

## 5.1.2. Per-protocol analyses of the primary outcome

Per-protocol analysis will also be performed by using GLMM model (as described in 5.1.1).

## 5.1.3. Covariate adjusted analysis of the primary outcome

An analysis of the primary outcome will be adjusted for, sex (binary), admission height(continuous), admission weight (continuous), admission age (continuous), admission IQ score (continuous), regular exercise time prior to admission(continuous) and admission medical usage (using medicine or not when enrolled, binary) of the primary outcome by GLMM model (as described in 5.1.1).

If the above GLMM model does not converge, GLMM model will be performed with less covariates until coverage.

Covariate adjusted analysis will be performed on both mITT and PP populations.

# **5.1.4.** Subgroup analyses of the primary outcome

Subgroup analyses will be performed for the primary outcome if each subgroup contains enough subject after stratification. We will stratify by sex (binary), categorized baseline medication usage (using medicine or not when enrolled, binary), qualified exercise days (less than 30/36/42/48 days, respectively, binary), categorized baseline exercise habit(binary), categorized baseline WFIRS score, and categorized baseline

SNAP score, respectively. (According to the scale rules, the continues variable will be transformed to the categorical variable.)

Subgroup analyses will be performed on both mITT and PP populations.

# 5.2. Secondary Outcome Analysis

All secondary outcomes will be analyzed as for a superiority designed trial and two-sided significance with alpha=5% and standard 95% CIs for the treatment differences in these outcomes between two groups will be calculated and presented. Secondary outcome analyses will be based on the mITT population unless specified.

The continuous outcome such as weight will be summarized using number of subjects (n), mean, standard deviation (SD), minimum, and maximum by treatment group, and will be analyzed by a GLMM model. Mean differences with 95% confidence intervals between two groups will be derived from the GLMM model.

All the secondary outcomes would be analyzed in the same tactics of primary outcome described above.

## 5.2.1. Handling of Missing data

Missing baseline covariates will be imputed using simple imputation methods in the covariate adjusted analysis based on the covariate distributions, should the missing values for a particular covariate be less than 5%. For a continuous variable, missing values will be imputed from random values from a normal distribution with mean and SD calculated from the available sample. For a categorical variable, missing values will be imputed from random values from a uniform distribution with probabilities P1,

P2, ..., and Pk from the sample. The seed to be used is 20211215.

# 6.General Considerations for Data Analyses

SAS (version 9.4) will be used to perform all data analyses and generate majority of data displays. STATA® (version 16.0) or R may also be used for some data analyses and generating statistical graphs.

#### 6.1. Other Data Summaries

Continuous variables will be summarized according to number of subjects without missing data (n), mean, standard deviation (SD), median range interquartile (IQR), minimum, and maximum. The confidence intervals will be reported on summaries of continuous effectiveness variables. Categorical variables will be summarized according to the absolute frequency and percentage of subjects (%) by category levels. The denominator for the percentages is the number of subjects in the treatment arm with data available, unless noted otherwise. Effect size ( $\eta$ <sup>2</sup>, eta-squared) would be estimated by SAS by PROC marco %effect\_size or by R software with effectsize package.

## 6.2. Graphical/Table Displays

Mean values for some continuous outcomes by treatment and visit will be plotted.

Table 1A Baseline characteristics of patients mITT Population

| Variable | Statistics | Treatment A (N=) | Treatment B (N=) |
|------------------------|------------|------------------|------------------|
| Age at baseline (year) | Mean(SD) | | |
| Height(cm) | Mean(SD) | | |
| Weight(kg) | Mean(SD) | | |

| Variable | Statistics | Treatment A (N=) | Treatment B (N=) |
|---|---|---|---|
| Using drug | Yes | | |
| | No | | |
| Gender | Female | | |
| | Male | | |
| SNAP scale score-INA-Doctor | Mean(SD) | | |
| SNAP scale score-HYP-Doctor | Mean(SD) | | |
| SNAP scale score-ODD-Doctor | Mean(SD) | | |
| SNAP scale score -INA -Parents | Mean(SD) | | |
| SNAP scale score-HYP-Parents | Mean(SD) | | |
| SNAP scale score-ODD-Parents | Mean(SD) | | |

Table 2: Summary statistics of primary and secondary outcomes: changes from baseline

| | | | Treatment A | Treatment B |
|---|---|---|---|---|
| Measurements | Visit | Statistics | (N=) | (N=) |
| SNAP scale score-<br>INA-Doctor | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| SNAP scale score-<br>HYP-Doctor | 3 months | n | | |
| | | Mean | | |

| | | | Treatment | Treatment |
|---|---|---|---|---|
| Measurements | Visit | Statistics | A<br>(N=) | B<br>(N=) |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| SNAP scale score-<br>ODD-Doctor | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| SNAP scale score -<br>INA -Parents | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |

| | | | Treatment | Treatment |
|---|---|---|---|---|
| | | | A | В |
| Measurements | Visit | Statistics | (N=) | (N=) |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| SNAP scale score-<br>HYP-Parents | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| SNAP scale score-<br>ODD-Parents | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |

| | | | Treatment | Treatment |
|---|---|---|---|---|
| Measurements | Visit | Statistics | A<br>(N=) | B<br>(N=) |
| Wicasurements | VISIT | Median | (11-) | (14-) |
| | | Maximum | | |
| D · | 2 41 | | | |
| Parent version of<br>Achenbach Child<br>Behavior Checklist<br>(CBCL) | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| Self-rated Strengths<br>and Difficulties<br>Questionnaire (SDQ) | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |

| | | | Treatment | Treatment |
|---|---|---|---|---|
| | | | A | В |
| Measurements | Visit | Statistics | (N=) | (N=) |
| | | Maximum | | |
| Weiss Functional<br>Impairment Rating<br>Scale (WFIRS) | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| Visual Perception-2nd edition (DTVP-2) | 3 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| Child Sensory<br>Integration Checklist | 3 months | n | | |

| | | | Treatment A | Treatment B |
|--------------|----------|------------|-------------|-------------|
| Measurements | Visit | Statistics | (N=) | (N=) |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |
| | 6 months | n | | |
| | | Mean | | |
| | | SD | | |
| | | Minimum | | |
| | | Median | | |
| | | Maximum | | |

Table 3.: Summary of mixed model analysis of primary and secondary outcomes

| | | n,mea | n (SD) | Mixed model an | alysis |
|---|---|---|---|---|---|
| Primary and secondary outcomes | Visit | Treatment A (N=306) | Treatment B (N=306) | Difference (95%CI) | p-value |
| SNAP scale score-INA-Doctor | 3 months | | | | |
| | 6 months | | | | |
| SNAP scale score-HYP-Doctor | 3 months | | | | |
| | 6 months | | | | |
| SNAP scale score-ODD-Doctor | 3 months | | | | |
| | 6 months | | | | |
| SNAP scale score -INA -Parents | 3 months | | | | |
| | 6 months | | | | |
| SNAP scale score-HYP-Parents | 3 months | | | | |
| | 6 months | | | | |
| SNAP scale score-ODD-Parents | 3 months | | | | |
| | 6 months | | | | |

| | | n,mean (SD) | | Mixed model analysis | |
|---|---|---|---|---|---|
| Primary and secondary outcomes | Visit | Treatment A (N=306) | Treatment B (N=306) | Difference (95%CI) | p-value |
| Parent version of Achenbach Child Behavior Checklist (CBCL) | 3 months | | | | |
| | 6 months | | | | |
| Self-rated Strengths and Difficulties Questionnaire (SDQ) | 3 months | | | | |
| | 6 months | | | | |
| Weiss Functional Impairment Rating Scale (WFIRS) | 3 months | | | | |
| | 6 months | | | | |
| Visual Perception-2nd edition (DTVP-2) | 3 months | | | | |
| | 6 months | | | | |
| Child Sensory Integration Checklist | 3 months | | | | |
| | 6 months | | | | |

Additional tables would be generated if more analysis were conducted.

# 7. Study variable list

| Variable | Туре |
|----------------|-------------|
| name | categorical |
| randomid | categorical |
| clinicalid | categorical |
| counselid | categorical |
| method | categorical |
| informaconsent | categorical |
| startdate | date |
| enddate | date |
| signature | categorical |
| inclusion1 | categorical |

| inclusion2 | categorical |
|---------------|-------------|
| inclusion3 | categorical |
| | _ |
| inclusion4 | categorical |
| inclusion5 | categorical |
| inclusion6 | categorical |
| metasiono | categorical |
| inclusion7 | categorical |
| inclusion8 | categorical |
| inclusion9 | categorical |
| exclusion1 | categorical |
| | S |
| exclusion2 | categorical |
| CACIUSIOII2 | categorical |
| exclusion3 | categorical |
| exclusion4 | categorical |
| exclusion5 | categorical |
| exclusion6 | categorical |
| exclusion7 | categorical |
| exclusion8 | categorical |
| firstcomplete | categorical |
| birthday | date |
| fathertel | categorical |
| mothertel | categorical |
| length | continuous |
| weight | continuous |
| peclass | continuous |
| oxtime | continuous |
| ropeskipping | continuous |

| slowrunning | continuous |
|-----------------------|-------------|
| quickrunning | continuous |
| pingpang | continuous |
| badminton | continuous |
| basketball | continuous |
| football | continuous |
| dancing | continuous |
| taekwondo | continuous |
| wushu | continuous |
| bicycle | continuous |
| otherpe | categorical |
| otherpe | categorical |
| medicalusage | categorical |
| medicalusagetime | continuous |
| TotalIQ | continuous |
| languageunderstanding | continuous |
| Preconception | continuous |
| remember | continuous |
| processspeed | continuous |
| DSNAP_INA | continuous |
| DSNAP_HYP | continuous |
| DSNAP_ODD | continuous |
| PSNAP_INA | continuous |
| PSNAP_HYP | continuous |
| PSNAP_ODD | continuous |
| DTVPGVP | continuous |
| DTVPMRP | continuous |
| DTVPVMI | continuous |
| PSDQmotion | continuous |
| PSDQbehavior | continuous |
| PSDQhyperactivity | continuous |
| PSDQcompany | continuous |
| PSDQsocial | continuous |
| PSDQhardrelationT | continuous |
| CSDQmotion | continuous |
| CSDQbehavior | continuous |
| CSDQhyperactivity | continuous |
| CSDQcompany | continuous |
| CSDQsocial | continuous |
| CSDQhardrelationT | continuous |
| Gantong1 | continuous |
| Gantong2 | continuous |
| <u> </u> | |

| 0 4 2 | |
|-----------------------------|-------------|
| Gantong3 | continuous |
| Gantong4 | continuous |
| Gantong5 | continuous |
| Gantong6 | continuous |
| Gantong7 | continuous |
| Gantong8 | continuous |
| Gantong9 | continuous |
| CBCL_1 | continuous |
| CBCL_2 | continuous |
| CBCL_3 | continuous |
| CBCL_4 | continuous |
| CBCL_5 | continuous |
| CBCL_6 | continuous |
| CBCL_7 | continuous |
| CBCL_8 | continuous |
| CBCL_9 | continuous |
| WEISSfamily | continuous |
| WEISSstudyschool | continuous |
| WEISSlifeskill | continuous |
| WEISSself | continuous |
| WEISSsocial | continuous |
| WEISSadventure | continuous |
| inhibitT | continuous |
| Self-monitor T | continuous |
| Shift T | continuous |
| Emotional Control T | continuous |
| Initiate T | continuous |
| Working memory T | continuous |
| Plan/Organize T | continuous |
| Task-monitor T | continuous |
| Organization of materials T | continuous |
| BRI T | continuous |
| ERI T | continuous |
| CRIT | continuous |
| GEC T | continuous |
| TCM shehong | continuous |
| TCM shetai | continuous |
| TCM mai | continuous |
| TCM total | continuous |
| testdate | date |
| complete | categorical |

| whostop | categorical |
|--------------------------|-------------|
| otherstop | categorical |
| stopreason | categorical |
| • | 5 |
| otherstopreason | categorical |
| AE | categorical |
| AEdetail | categorical |
| AEdeal | categorical |
| usemedicine | categorical |
| | - |
| usemedicinedose | continuous |
| otherusemedicinedose | categorical |
| TotalIQ 3m | continuous |
| languageunderstanding_3m | continuous |
| Preconception_3m | continuous |
| remember_3m | continuous |
| processspeed_3m | continuous |
| DSNAP_INA_3m | continuous |
| DSNAP_HYP_3m | continuous |
| DSNAP_ODD_3m | continuous |
| PSNAP_INA_3m | continuous |
| PSNAP_HYP_3m | continuous |
| PSNAP_ODD_3m | continuous |
| DTVPGVP_3m | continuous |
| DTVPMRP_3m | continuous |
| DTVPVMI_3m | continuous |
| PSDQmotion_3m | continuous |
| PSDQbehavior_3m | continuous |
| PSDQhyperactivity_3m | continuous |
| PSDQcompany_3m | continuous |
| PSDQsocial_3m | continuous |
| PSDQhardrelationT_3m | continuous |
| CSDQmotion_3m | continuous |
| CSDQbehavior_3m | continuous |
| CSDQhyperactivity_3m | continuous |
| CSDQcompany_3m | continuous |

| CSDQsocial 3m | continuous |
|--------------------------------|------------|
| CSDQhardrelationT 3m | continuous |
| Gantong1 3m | continuous |
| Gantong2_3m | continuous |
| Gantong3 3m | continuous |
| Gantong4 3m | continuous |
| Gantong5 3m | continuous |
| Gantong6 3m | continuous |
| Gantong7 3m | continuous |
| Gantong8 3m | continuous |
| Gantong9 3m | continuous |
| CBCL 1 3m | continuous |
| | continuous |
| CBCL_2_3m | |
| CBCL_3_3m | continuous |
| CBCL_4_3m | continuous |
| CBCL_5_3m | continuous |
| CBCL_6_3m | continuous |
| CBCL_7_3m | continuous |
| CBCL_8_3m | continuous |
| CBCL_9_3m | continuous |
| WEISSfamily_3m | continuous |
| WEISSstudyschool_3m | continuous |
| WEISSlifeskill_3m | continuous |
| WEISSself_3m | continuous |
| WEISSsocial_3m | continuous |
| WEISSadventure_3m | continuous |
| inhibitT_3m | continuous |
| Self-monitor T_3m | continuous |
| Shift T_3m | continuous |
| Emotional Control T_3m | continuous |
| Initiate T_3m | continuous |
| Working memory T_3m | continuous |
| Plan/Organize T_3m | continuous |
| Task-monitor T_3m | continuous |
| Organization of materials T_3m | continuous |
| BRI T_3m | continuous |
| ERI T_3m | continuous |
| CRI T_3m | continuous |
| GEC T_3m | continuous |
| TCM_shehong_3m | continuous |
| TCM_shetai_3m | continuous |
| TCM_mai_3m | continuous |

| TCM total 3m | continuous |
|--------------------------------------|--------------------------|
| testdate | date |
| complete | categorical |
| whostop | categorical |
| otherstop | categorical |
| stopreason | categorical |
| otherstopreason | categorical |
| AE | categorical |
| AEdetail | categorical |
| AEdeal | categorical |
| usemedicine | categorical |
| usemedicinedose | continuous |
| otherusemedicinedose | categorical |
| TotalIQ_6m | continuous |
| languageunderstanding_6m | continuous |
| Preconception_6m | continuous |
| remember_6m | continuous |
| processspeed_6m | continuous |
| DSNAP_INA_6m | continuous |
| DSNAP_HYP_6m | continuous |
| DSNAP_ODD_6m | continuous |
| PSNAP_INA_6m | continuous |
| PSNAP_HYP_6m | continuous |
| PSNAP_ODD_6m | continuous |
| DTVPGVP_6m | continuous |
| DTVPMRP_6m | continuous |
| DTVPVMI_6m | continuous |
| I DODO | 1 |
| PSDQmotion_6m | continuous |
| PSDQmotion_6m PSDQbehavior_6m | continuous continuous |
| PSDQbehavior_6m | continuous |
| PSDQbehavior_6m PSDQhyperactivity_6m | continuous<br>continuous |

| GGD 0 | |
|--------------------------------|------------|
| CSDQmotion_6m | continuous |
| CSDQbehavior_6m | continuous |
| CSDQhyperactivity_6m | continuous |
| CSDQcompany_6m | continuous |
| CSDQsocial_6m | continuous |
| CSDQhardrelationT_6m | continuous |
| Gantong1_6m | continuous |
| Gantong2_6m | continuous |
| Gantong3_6m | continuous |
| Gantong4_6m | continuous |
| Gantong5_6m | continuous |
| Gantong6_6m | continuous |
| Gantong7_6m | continuous |
| Gantong8_6m | continuous |
| Gantong9_6m | continuous |
| CBCL_1_6m | continuous |
| CBCL_2_6m | continuous |
| CBCL_3_6m | continuous |
| CBCL_4_6m | continuous |
| CBCL_5_6m | continuous |
| CBCL_6_6m | continuous |
| CBCL_7_6m | continuous |
| CBCL_8_6m | continuous |
| CBCL_9_6m | continuous |
| WEISSfamily_6m | continuous |
| WEISSstudyschool_6m | continuous |
| WEISSlifeskill_6m | continuous |
| WEISSself_6m | continuous |
| WEISSsocial_6m | continuous |
| WEISSadventure_6m | continuous |
| inhibitT_6m | continuous |
| Self-monitor T 6m | continuous |
| Shift T_6m | continuous |
| Emotional Control T_6m | continuous |
| Initiate T 6m | continuous |
| Working memory T 6m | continuous |
| Plan/Organize T 6m | continuous |
| Task-monitor T 6m | continuous |
| Organization of materials T_6m | continuous |
| BRI T_6m | continuous |
| ERI T_6m | continuous |
| CRI T_6m | continuous |

| GEC T_6m | continuous |
|----------------|------------|
| TCM_shehong_6m | continuous |
| TCM_shetai_6m | continuous |
| TCM_mai_6m | continuous |
| TCM_total_6m | continuous |

# 8.Reference

[1] Jin W, Du Y, Zhong X, David C. Prevalence and contributing factors to attention deficit hyperactivity disorder: a study of five- to fifteen-year-old children in Zhabei District, Shanghai. Asia Pac Psychiatry. 2014;6:397-404.